CLINICAL TRIAL: NCT03751241
Title: Evaluation of Reading Quality in Three Different Patient Groups (Extended Range Of Vision vs Minimonovision vs Single Focus Distance Vision)
Brief Title: Reading Quality in Three Different Patient Groups
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Eyetracker
Record Dates: First submitted 2018-11-21; First posted 2018-11-23 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Pseudophakia
Keywords: Pseudophakia; Reading speed
MeSH Terms: conditions — Pseudophakia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraocular lens types (Experimental): Patients with different types of IOLs (EROV, monofocal, minimonovision) are tested for their reading quality using the EyeTracker device
  Interventions: Device: EyeTracker

INTERVENTIONS:
Device: EyeTracker — The EyeTracker is used to determine reading quality of patients with different intraocular lens types (EROV, monofocal, minimonovision)

SUMMARY:
Influence of different ophthalmic conditions after cataract surgery (extended range of vision IOL (EROV) with micromonovision, minimonovision with standard IOL and single focus distance vision with standard IOL) on reading quality.

DETAILED DESCRIPTION:
Reading is a complex function. It requires a proper retinal image that is received by the brain. There it is analyzed for letter and word recognition and then the semantics is detected. Reading speed slows down when letters are blurred, or do not have enough contrast or luminance or when binocular fusion is hampered. It also slows down when the understanding is difficult, which is why reading one's mother tongue generally is faster than reading a foreign language. Reading skill is therefore influenced by visuo-motor and cognitive (i.e. linguistic, personality, learning, ageing) factors. Reading ability is currently evaluated using various reading tests, which usually have long paragraphs with small print and shorter ones with larger print, to allow determination of reading acuity. To evaluate sustained reading performance, and reading speed, the International Reading Speed Texts (IReST) which contain longer paragraphs with continuous text of fixed size, have been developed. Although clinical reading tests are thoroughly standardized, a significant inter-individual variation in reading speed exists, as a result of the high influence of cognitive factors. When reading, sensorimotor coordination must happen to make a sequence of fixations and saccades so that new information falls onto the fovea. Eye movement efficiency develops almost in parallel with reading ability, in terms of speed and accuracy, as the child progresses from a beginner to a proficient adult reader. Less skilled readers (e.g. children with reading difficulties) typically make more fixations of longer duration and shorter saccades than skilled readers. For an adult reader mean fixation duration is around 220 to 250 ms. However, fixations of variable durations (from 100 ms to over 500 ms) are recorded during a reading session. Although the distribution of fixation durations varies among individuals, due to differences in reading skill, age and other cognitive factors, it is never normal; it always exhibits a pronounced right tail, i.e. an increased frequency of long fixations. Such distributions can be fitted with an ex-Gaussian function, a convolution of Gaussian (normal) and exponential functions, which could provide more efficient analysis. The team in university of Crete recently showed that pre-retinal factors (e.g. text contrast and luminance) influence the mean of the normal distribution, while cognitive factors affect the number of fixations and the mean of the exponential distribution of fixation duration, due to an increased frequency of long fixations. Moreover, inter-individual variation was significantly improved when analysis was performed separately for visuo-motor vs. cognitive components, with most of variability being attributed to the mean of the exponential distribution.

To evaluate functional vision in "simultaneous-image' correction and more specifically visual performance at near, a functional outcome, such as reading speed and ocular fixation times during sustained reading, should be measured. Such recordings could then answer the question how the binocular improvement in reading depends on the difference in acuity between the eyes and the analysis suggested above could help us to distinguish sensory vs. motor components especially in patients with reduced contrast sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 and older
* Written informed consent
* Extended range of vision group: Patients with EROV intraocular lenses and a best-corrected Snellen VA above 0.7 in the weaker eye. Furthermore, the VA of the better eye has to be at least 0.8 (uncorrected visual acuity) and the difference between the eyes should be between 0.5D and 1D)
* Minimonovision standard IOL group: Patients with monofocal intraocular lenses and a best-corrected Snellen VA above 0.7 in the weaker eye. Furthermore, the VA of the better eye has to be at least 0.8 (uncorrected visual acuity) and the difference between the eyes should be between 0.75D and 1.50D)
* Single focus distance vision group: Patients with monofocal intraocular lenses and a best-corrected Snellen VA above 0.7 in the weaker eye. Furthermore, the VA of the better eye has to be at least 0.8 (uncorrected visual acuity) and both eyes should have a spherical equivalent between +0.25D and -0.5D
* Maximum of allowed Cylinder: +0.75D
* Fluent in German

Exclusion Criteria:

* Opacities, such as corneal scars
* In case of pregnancy (pregnancy test will be taken preoperatively in women of reproductive age)

Ages: 21 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Reading speed | 12 months
  Reading speed in the 3 different IOL groups (EROV, monofocal, minimonovision) will be assessed using the EyeTracker device. Patients are asked to read 4 texts with different contrast levels. The faster the patients can read the texts, the better the outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided